CLINICAL TRIAL: NCT00414323
Title: Evaluation of the Effects of Duloxetine on Norepinephrine Transporter Inhibition in Healthy Subjects
Brief Title: Evaluation of the Effects of Duloxetine on Norepinephrine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 9547; F1J-MC-HMEU
Record Dates: First submitted 2006-12-15; First posted 2006-12-21 (Estimated); Last update posted 2007-06-12 (Estimated); Status verified 2007-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride; Escitalopram

INTERVENTIONS:
Drug: Duloxetine
Drug: Escitalopram
Drug: Placebo

SUMMARY:
The purpose of this study is to evaluate how taking duloxetine 60mg every day affects the transfer of two normal body chemicals, 3,4-dihydroxyphenylglycol (DHPG) and norepinephrine (NE), across cells in blood and cerebrospinal fluid.

ELIGIBILITY:
Healthy subjects between the ages of 18-65 years are nonsmokers or are willing to refrain from smoking and are not taking concomitant medications which may inhibit or induce CYP1A2 or CYPD6 or is an MAOI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-11; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Concentrations of DHPG and NE in plasma (in sitting and standing positions), urine, and CSF after multiple daily doses (steady state).

SECONDARY OUTCOMES:
Effect of duloxetine versus escitalopram on ex vivo reuptake inhibition of NE and F-hydroxytryptamine (5-HT) in serum and relationship to exposure.
Effect of duloxetine versus escitalopram on heart rate variability.
Ratio of duloxetine exposure in plasma to CSF at steady state.
Relationship between DHPG and NE concentrations and duloxetine exposure in CSF and plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas